CLINICAL TRIAL: NCT01307774
Title: Survey of Predictors of HPV Vaccination Among Parents of Rural Adolescent Girls in Mysore, India
Brief Title: Survey of Predictors of Human Papillomavirus (HPV) Vaccination Among Parents of Rural Adolescent Girls in Mysore, India
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Purnima Madhivanan (Other)
Collaborators: Florida International University (Other)
Responsible Party: Sponsor-Investigator, Purnima Madhivanan, Principal Investigator, Public Health Research Institute, India
Organization: Public Health Research Institute, India (Other)
Other Study IDs: IISP38250
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Human Papillomavirus; Cervical Cancer
Keywords: parental acceptability of HPV vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To conduct a quantitative survey to measure knowledge about Human papillomavirus (HPV) and cervical cancer, and HPV vaccine acceptability among parents of rural adolescent girls in Mysore District, India.

Hypothesis: General knowledge and attitudes about the severity and treat ability of cancer will predict acceptability of HPV vaccination among parents of rural adolescent girls in Mysore, India.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* parent of an adolescent girl (10 -15 years of age)
* able to speak English or Kannada
* willing to undergo informed consent process

Exclusion Criteria:

* Does not have the capacity to undergo informed consent process

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will survey attitudes of parents of adolescent girls attending 10 schools in rural Mysore Taluk in Mysore District.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Parental Acceptability of HPV vaccine | One year

SECONDARY OUTCOMES:
Knowledge about HPV and Cervical Cancer | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Madhivanan, MBBS, PhD, Principal Investigator — Public Health Research Institute of India
Locations (1):
- Public Health Research Institute of India, Mysore, Karnataka, India

REFERENCES:
- [Background] Madhivanan P, Krupp K, Yashodha MN, Marlow L, Klausner JD, Reingold AL. Attitudes toward HPV vaccination among parents of adolescent girls in Mysore, India. Vaccine. 2009 Aug 20;27(38):5203-8. doi: 10.1016/j.vaccine.2009.06.073. Epub 2009 Jul 9. PMID 19596420
- [Background] Krupp K, Marlow LA, Kielmann K, Doddaiah N, Mysore S, Reingold AL, Madhivanan P. Factors associated with intention-to-recommend human papillomavirus vaccination among physicians in Mysore, India. J Adolesc Health. 2010 Apr;46(4):379-84. doi: 10.1016/j.jadohealth.2009.10.001. Epub 2009 Nov 24. PMID 20307828